CLINICAL TRIAL: NCT02535221
Title: Randomized Trial of Neoadjuvant Endocrine Therapy Versus Chemotherapy in Premenopausal Patients With Estrogen Receptor-Positive HER2 Negative Breast Cancer
Brief Title: Neoadjuvant Endocrine Therapy Versus Chemotherapy in Premenopausal Patients With ER+ & HER2- Breast Cancer
Status: Recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: Peking University (Other)
Responsible Party: Principal Investigator, Tao OUYANG, Chairman of Breast Center of Peking University Cancer Hospital, Peking University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: BCP12
Record Dates: First submitted 2015-06-09; First posted 2015-08-28 (Estimated); Last update posted 2021-11-29 (Actual); Status verified 2021-11

CONDITIONS: Breast Cancer
Keywords: Premenopausal Patients; Estrogen Receptor-Positive HER2 negative
MeSH Terms: conditions — Breast Neoplasms | interventions — Drug Therapy

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Endocrine therapy; (Experimental): Interventions：Goserelin+TAM+AI：Goserelin 3.6mg subcutaneous injection per 4 weeks, for 16-20weeks. TAM 10mg oral twice a day for the first four weeks(to wait the Goserelin start to work in body) than change to AI 1mg oral once a day with Goserelin for the next 12-16 weeks.
  Interventions: Drug: Goserelin+TAM+AI
- Chemotherapy (Active Comparator): Interventions：Epirubicin+CTX+5-Fu：Epirubicin(80-100 mg/m2 Q21 days) + CTX(600 mg/m2 Q 21days) + 5-Fu (600 mg/m2 Q21 days or 200 mg/m2 •day from Day1 to day 21) for four to six cycles.
  Interventions: Drug: Epirubicin+CTX+5-Fu

INTERVENTIONS:
Drug: Goserelin+TAM+AI — Goserelin 3.6mg subcutaneous injection per 4 weeks, for 16-20weeks. TAM 10mg oral twice a day for the first four weeks(to wait the Goserelin start to work in body) than change to AI 1mg oral once a day with Goserelin for the next 12-16 weeks.
  Other Names: Endocrine therapy
  Arms: Endocrine therapy;
Drug: Epirubicin+CTX+5-Fu — Epirubicin(80-100 mg/m2 Q21 days) + CTX(600 mg/m2 Q 21days) + 5-Fu (600 mg/m2 Q21 days or 200 mg/m2 •day from Day1 to day 21) for four to six cycles.
  Other Names: Chemotherapy
  Arms: Chemotherapy

SUMMARY:
This study proposes to prove that the efficacy of adjuvant endocrine therapy for the premenopausal HR positive breast cancer patients is non-inferiority to adjuvant chemotherapy assessed by ultrasound response rate.

ELIGIBILITY:
Inclusion Criteria:

* 35 years old <age≤55 years old, in premenopausal status(with the judgement by researchers when the patients are recruited) Histologically confirmed primary invasive breast cancer
* Stage: T2N0M0(cT>2cm, SLNB negative), hard to proceed the breast conserving surgery(not feasible or may affect the appearance of breast)
* Histologically confirmed HR+ (ER or PR positive, and >50% cell in IHC) HER2 negative breast cancer by pathological evaluation
* No other previous treatment for primary breast cancer
* Without other tumor or unstable complication or uncontrolled infection
* No contradiction for the third generation AIs, LHRHa, chemotherapy
* Attend the study voluntarily, sign the informed consent.

Exclusion Criteria:

* Metastasis disease by pathological or radiological diagnosis
* the history of other tumor
* contradiction for the third generation AIs, LHRHa, chemotherapy
* Contradiction for adjuvant chemotherapy: serious cardiology or cerebral vessel disease, liver or kidney disfunction, blood system disease, the other situation or complication that are not suitable or cannot adaptable for chemotherapy
* Contradiction for proceeding surgery: contradiction for anesthesia, large lesion,T4, lymph node positive
* other situation not suitable for the research: psychological disease, mental disorder, social problem, geographic problem
* have been attendance in other anti-tumor treatment or other clinical trials 8) reject to attend the study

Ages: 35 Years to 55 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 234 (Estimated)
Dates: Start 2015-07-29 (Actual); Primary Completion 2026-06-30 (Estimated); Study Completion 2026-12-31 (Estimated)

PRIMARY OUTCOMES:
ultrasound response rate | within 2 weeks before surgery

SECONDARY OUTCOMES:
pathological response rate(Miller & Payne standard) | with 2 weeks after surgery

CONTACTS AND LOCATIONS:
Overall Officials: Tao Ouyang, MD, Study Chair — Peking University Cancer Hospital & Institute
Locations (1):
- Beijing Cancer Hospital Breast Center, Beijing, China

REFERENCES:
- [Derived] Gu C, He Y, Zhang N, Liu Y, Li J, Wang T, Fan T, Fan Z, Ouyang T. A Non-Inferior Randomized Trial of Neoadjuvant Endocrine Therapy Compared to Neoadjuvant Chemotherapy in Premenopausal Patients With Hormone-Responsive and HER2-Negative Lymph Node-Negative Breast Cancer. Cancer Control. 2025 Jan-Dec;32:10732748251339958. doi: 10.1177/10732748251339958. Epub 2025 May 7. PMID 40331570